CLINICAL TRIAL: NCT00240006
Title: An Open Label, Prospective Parallel Cohort Study Comparing A 90-day Copaxone® Adherence Enhancement Program Among Persons With Multiple Sclerosis Who Participate in Shared Solutions® Alone or in Partnership With Their MS Center
Brief Title: A Study Comparing Shared Solutions® Plus MS Center Support Versus Shared Solutions® Alone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Neuroscience, Inc. (Industry)
Responsible Party: Siyu Liu, Senior Director of Pan Am Clinical Operations, Teva Neuroscience
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PM024
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Copaxone®; Shared Solutions®
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Shared Solutions®
  Interventions: Procedure: Shared Solutions® plus MS Center v. Shared Solutions®
- 2 (Experimental): Shared Solutions® and MS Center/Office Practice Partnership
  Interventions: Procedure: Shared Solutions® plus MS Center v. Shared Solutions®

INTERVENTIONS:
Procedure: Shared Solutions® plus MS Center v. Shared Solutions® — Copaxone

SUMMARY:
To compare the effectiveness of a 90-day Copaxone® adherence enhancement program for a sample of MS patients who are at high risk of nonadherence and receive support from Shared Solutions® and their MS Center versus those who receive support only from Shared Solutions®.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18 years of age or older.
2. Diagnosed with Relapsing Remitting Multiple Sclerosis (relapses accepted).
3. Beginning or restarting therapy with Glatiramer Acetate (Copaxone®).
4. Willing and able to complete all procedures and evaluations related to the study.
5. Willing to provide informed consent.

Exclusion Criteria:

1. Taking any other immunomodulatory or immunosuppressant therapy in conjunction with Copaxone®.
2. Has a significant medical illness other than MS that may interfere with the assessment of endpoints or the subject's participation in the trial for the full duration of the study.
3. Any situation that the investigator or nurse (if not the investigator) feel may interfere with participation in the study.
4. Pregnant or trying to become pregnant, or breast feeding during the study.
5. Previously participated in this study or another clinical research study in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Adherence rate of Copaxone therapy by procedural intervention | 90 days

SECONDARY OUTCOMES:
Compliance of treatment, positive experience of treatment, levels of depression, proportion of time spent, self injection competency ratings, and the risk of non-adherence/non-compliance | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: MerriKay Oleen-Burkey, Ph.D., Study Director — Teva Neuroscience, Inc.